CLINICAL TRIAL: NCT02465268
Title: ATTAC-II: A Phase II Randomized, Blinded, and Placebo-controlled Trial of CMV RNA-Pulsed Dendritic Cells With Tetanus-Diphtheria Toxoid Vaccine in Patients With Newly-Diagnosed Glioblastoma
Brief Title: Vaccine Therapy for the Treatment of Newly Diagnosed Glioblastoma Multiforme
Acronym: ATTAC-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201400697-N; R01CA175517 (NIH); OCR14127 (Other: Universiy of Florida)
Record Dates: First submitted 2015-05-27; First posted 2015-06-08 (Estimated); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Glioblastoma Multiforme; Glioblastoma; Malignant Glioma; Astrocytoma, Grade IV; GBM
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Sodium Chloride; Tetanus Toxoid; Diphtheria Toxoid; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: pp65-shLAMP DC with GM-CSF and Td (Experimental): Given under the skin at day 22-24 after the first temozolomide cycle then at 2 week intervals. Doses 4-10 will be given on day 22-24 of each temozolomide cycle. Doses will continue until a total of 10 or until progression or unacceptable toxicity.
  Interventions: Biological: pp65-shLAMP DC with GM-CSF; Drug: Td
- Arm 2: pp65-flLAMP DC with GM-CSF and Td (Experimental): Given under the skin at day 22-24 after the first temozolomide cycle then at 2 week intervals. Doses 4-10 will be given on day 22-24 of each temozolomide cycle. Doses will continue until a total of 10 or until progression or unacceptable toxicity.
  Interventions: Drug: Td; Biological: pp65-flLAMP DC with GM-CSF
- Arm 3: unpulsed PBMC and Saline (Placebo Comparator): Given under the skin at day 22-24 after the first temozolomide cycle then at 2 week intervals. Doses 4-10 will be given on day 22-24 of each temozolomide cycle. Doses will continue until a total of 10 or until progression or unacceptable toxicity.
  Interventions: Biological: unpulsed PBMC and saline; Drug: Saline

INTERVENTIONS:
Biological: pp65-shLAMP DC with GM-CSF
  Other Names: pp65-shLAMP mRNA DCs with GM-CSF
  Arms: Arm 1: pp65-shLAMP DC with GM-CSF and Td
Biological: unpulsed PBMC and saline
  Other Names: Peripheral Blood Mononuclear Cells
  Arms: Arm 3: unpulsed PBMC and Saline
Drug: Td — All subjects will receive a Td booster before study drug dose #1. Subjects in the experimental arms will receive Td skin prep before study drug doses #3, #6, and #9.
  Other Names: Tetanus and Diphtheria Toxoid
  Arms: Arm 1: pp65-shLAMP DC with GM-CSF and Td; Arm 2: pp65-flLAMP DC with GM-CSF and Td
Drug: Saline
  Other Names: Normal Saline
  Arms: Arm 3: unpulsed PBMC and Saline
Biological: pp65-flLAMP DC with GM-CSF
  Other Names: pp65-flLAMP mRNA DCs with GM-CSF
  Arms: Arm 2: pp65-flLAMP DC with GM-CSF and Td

SUMMARY:
The purpose of this research study is to determine if an investigational dendritic cell vaccine, called pp65 DC, is effective for the treatment of a specific type of brain tumor called glioblastoma (GBM) when given with stronger doses of routine chemotherapy.

DETAILED DESCRIPTION:
Dendritic cells (DC) are involved in activating, or turning-on, your body's immune system. Your immune system helps guard your body from germs, viruses, and other threats. Although dendritic cells are very strong, the number of them in the body is not high enough to cause a powerful immune response; therefore, more DC are made in a laboratory with cells collected from an individual's blood.

In this study, we will make a vaccine that we hope will educate immune cells to target the pp65 antigen, a type of immune marker in GBM, thus resulting in what we call the pp65 DC vaccine. Use of a vaccine that activates your immune system is a type of immunotherapy. It is hoped that by giving the pp65 DC vaccine as a shot under the skin, the immune system will be activated to attack tumor cells in the brain while leaving normal cells alone.

To see if the pp65 DC vaccine is effective for the treatment of GBM, subjects will be assigned to different treatment groups. Two groups of subjects will receive the pp65 DC vaccine and one group will receive a placebo.

ELIGIBILITY:
Abbreviated Inclusion Criteria:

To be assessed at study enrollment prior to standard of care chemo-radiation therapy:

* Age ≥ 18 years.
* Histopathologically proven newly-diagnosed de novo GBM (WHO Grade IV glioma)
* The tumor must have a supratentorial component.
* Must have undergone definitive surgical resection of tumor with less than approximately 3cm x 3cm residual enhancing tumor as product of longest perpendicular planes by MRI.
* Recovery from the effects of surgery, postoperative infection, and other complications.
* Diagnostic contrast-enhanced MRI or CT scan of the brain preoperatively and postoperatively.
* Karnofsky Performance Status of ≥ 70.
* Signed informed consent.
* For females of childbearing potential, negative serum pregnancy test.
* Women of childbearing potential and male participants must be willing to practice adequate contraception throughout the study and for at least 24 weeks after the last dose of study drug.

To be assessed prior to initiation of adjuvant TMZ:

* Must have completed RT (targeted total dose of 59.4-60.0 Gy over ≤ 7 weeks) and concomitant TMZ (targeted dose of 75mg/m2/d for ≤ 49 days) therapy without significant toxicity that persisted over 4 weeks.
* History & physical with neurologic examination prior to initiation of adjuvant TMZ.
* For patients receiving steroids, daily dose must be ≤ 4 mg.
* CBC with differential with adequate bone marrow function.
* Adequate renal function.
* Adequate hepatic function.

Abbreviated Exclusion Criteria:

To be verified in order to randomize subject:

* Prior invasive malignancy unless disease free for ≥ 3 years.
* Metastases detected below the tentorium or beyond the cranial vault and leptomeningeal involvement.
* Recurrent or multifocal malignant gliomas.
* HIV, Hepatitis B, or Hepatitis C seropositive.
* Known active infection or immunosuppressive disease.
* Prior chemotherapy or radiosensitizers (including Gliadel wafers) for cancers of the head and neck region.
* Prior radiotherapy to the head or neck, resulting in overlap of radiation fields.
* Severe, active co-morbidity.
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception for the entire study period.
* Pregnant or lactating women.
* Prior allergic reaction to temozolomide, GM-CSF or Td.
* Prior history of brachial neuritis or Guillain-Barré syndrome.
* Patients treated on any other therapeutic clinical protocols within 30 days prior to study entry.

To be assessed prior to initiation of adjuvant TMZ:

* Did not start radiation therapy and temozolomide within 7 weeks of surgery.
* Progression of disease as defined by modified RANO criteria.
* More than 45 days after completion of radiation therapy and temozolomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2016-08-09 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duane Mitchell, MD, PhD, Study Chair — University of Florida; Maryam Rahman, MD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Orlando Health, Orlando, Florida
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 175 participants were enrolled (consented) between 8/9/2016 and 10/5/2022.
Pre-assignment Details: Participants were evaluated for inclusion. 17 were determined not eligible and 4 participants withdrew. 154 participants were randomized with an allocation ratio of 1:1:1 into one of three arms: 1) Arm 1: pp65-shLAMP mRNA DCs with GM-CSF 150 µg (Td skin prep); 2) Arm 2: pp65-flLAMP mRNA DCs with GM-CSF 150 µg (Td skin prep); or 3) Arm 3: Unpulsed PBMCs (saline skin prep).
Groups:
- pp65-shLAMP DC With GM-CSF and Td (Arm 1): Prior to leukapheresis, patients will be randomized to receive one of three treatment regimens with dose-intensified TMZ treatment at 100 mg/m2/day for 21 days with an allocation ratio of 1:1:1 into one of three arms.
  Experimental Arm 1 pp65-shLAMP DC with GM-CSF and Td
  DC vaccines are given under the skin at day 22-24 after the first temozolomide cycle then at 2-week intervals. Doses 4-10 will be given on day 22-24 of each temozolomide cycle. Doses will continue until a total of 10 or until progression or unacceptable toxicity.
  Td: All subjects will receive a Td booster before study drug dose #1. Subjects in the experimental arms will receive Td skin prep before study drug doses #3, #6, and #9.
- pp65-flLAMP DC With GM-CSF and Td (Arm 2): Prior to leukapheresis, patients will be randomized to receive one of three treatment regimens with dose-intensified TMZ treatment at 100 mg/m2/day for 21 days with an allocation ratio of 1:1:1 into one of three arms.
  Experimental Arm 2 pp65-flLAMP DC with GM-CSF and Td
  DC vaccines are given under the skin at day 22-24 after the first temozolomide cycle then at 2-week intervals. Doses 4-10 will be given on day 22-24 of each temozolomide cycle. Doses will continue until a total of 10 or until progression or unacceptable toxicity.
  Td: All subjects will receive a Td booster before study drug dose #1. Subjects in the experimental arms will receive Td skin prep before study drug doses #3, #6, and #9.
- Unpulsed PBMC and Saline (Arm 3): The control group was Arm 3, Unpulsed PBMCs (saline skin prep)
  Prior to leukapheresis, patients will be randomized to receive one of three treatment regimens with dose-intensified TMZ treatment at 100 mg/m2/day for 21 days with an allocation ratio of 1:1:1 into one of three arms.
Period: Overall Study
Arm/Group | pp65-shLAMP DC With GM-CSF and Td (Arm 1) | pp65-flLAMP DC With GM-CSF and Td (Arm 2) | Unpulsed PBMC and Saline (Arm 3)
Started | 52 | 50 | 52
Completed | 36 | 34 | 41
Not Completed | 16 | 16 | 11
Not completed — Withdrawal by Subject | 4 | 3 | 1
Not completed — Not evaluable per protocol criteria | 3 | 2 | 1
Not completed — did not meet eligibility prior to Cycle #1 | 8 | 9 | 9
Not completed — Study drug did not pass QA/QC | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one DC vaccine were included in the modified intent to treat analysis.
Groups:
- pp65-shLAMP DC With GM-CSF and Td (Arm 1): The active treatment group were Arms 1 and 2
  Arm 1: pp65-shLAMP mRNA DCs with GM-CSF 150 µg (Td skin prep)
  Prior to leukapheresis, patients will be randomized to receive one of three treatment regimens with dose-intensified TMZ treatment at 100 mg/m2/day for 21 days with an allocation ratio of 1:1:1 into one of three arms.
- pp65-flLAMP DC With GM-CSF and Td (Arm 2): The active treatment group were Arms 1 and 2
  Arm 2: pp65-flLAMP mRNA DCs with GM-CSF 150 µg (Td skin prep)
  Prior to leukapheresis, patients will be randomized to receive one of three treatment regimens with dose-intensified TMZ treatment at 100 mg/m2/day for 21 days with an allocation ratio of 1:1:1 into one of three arms.
- Total: Total of all reporting groups
Arm/Group | pp65-shLAMP DC With GM-CSF and Td (Arm 1) | pp65-flLAMP DC With GM-CSF and Td (Arm 2) | Unpulsed PBMC and Saline (Arm 3) | Total
Number analyzed (Participants) | 36 | 34 | 41 | 111
Age, Continuous [Median (Full Range); unit: years] | 61.0 [32.0 to 75.0] | 56.0 [21.0 to 79.0] | 59.0 [27.0 to 80.0] | 58.0 [21.0 to 80.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 13 | 30
  Male | 28 | 25 | 28 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 3
  Not Hispanic or Latino | 34 | 34 | 35 | 103
  Unknown or Not Reported | 2 | 0 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 4
  White | 32 | 32 | 36 | 100
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 36 | 34 | 41 | 111

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Overall Survival (OS) Between the Active Treatment Group (Arms 1 and 2) and the Control Group (Arm 3)
Description: Kaplan-Meier survival curves and the log rank test will be used to characterize and compare OS in patients who received pp65-LAMP mRNA DC vaccine (Arms 1 and 2) and in control patients (Arm 3). OS will be defined as the time between first vaccination and death and will be censored at the last follow-up if death has not occurred.
Time Frame: From date of first vaccine until the date of death, up to 48 months
Population: Survival in Patients receiving vaccine vs placebo.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- pp65-shLAMP DC With GM-CSF and Td (Arm 1); pp65-flLAMP DC With GM-CSF and Td (Arm 2): Given under the skin at day 22-24 after the first temozolomide cycle then at 2 week intervals. Doses 4-10 will be given on day 22-24 of each temozolomide cycle. Doses will continue until a total of 10 or until progression or unacceptable toxicity.
  pp65-shLAMP DC with GM-CSF (Arm 1) pp65-flLAMP DC with GM-CSF (Arm 2)
  Td: All subjects will receive a Td booster before study drug dose #1. Subjects in the experimental arms will receive Td skin prep before study drug doses #3, #6, and #9.
- Unpulsed PBMC and Saline (Arm 3): Given under the skin at day 22-24 after the first temozolomide cycle then at 2 week intervals. Doses 4-10 will be given on day 22-24 of each temozolomide cycle. Doses will continue until a total of 10 or until progression or unacceptable toxicity.
  unpulsed PBMC and saline
  Saline
Arm/Group | pp65-shLAMP DC With GM-CSF and Td (Arm 1) | pp65-flLAMP DC With GM-CSF and Td (Arm 2) | Unpulsed PBMC and Saline (Arm 3)
Number analyzed (Participants) | 36 | 34 | 41
months | 16.9 [12.7 to 22.8] | 16.2 [13.8 to 19.2] | 20.6 [15.4 to 30.2]
Statistical Analysis 1: Comparison: pp65-shLAMP DC With GM-CSF and Td (Arm 1) vs Unpulsed PBMC and Saline (Arm 3); Test type: Superiority; p = 0.196, Log Rank; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.77 to 2.16]
Statistical Analysis 2: Comparison: pp65-flLAMP DC With GM-CSF and Td (Arm 2) vs Unpulsed PBMC and Saline (Arm 3); Test type: Superiority; p = 0.196, Log Rank; Hazard Ratio (HR) = 1.63, 95% CI 2-sided [0.99 to 2.70]

2. Secondary Outcome: Comparison of Progression-free Survival Between the Active Treatment Group (Arms 1 and 2 Combined) and the Control Group (Arm 3)
Description: Calculated as dated of first vaccine to date first progression/recurrence or death. Kaplan-Meier survival curves and the log rank test will be used to characterize and compare PFS in patients who received pp65-LAMP mRNA DC vaccine (Arms 1 and 2) and in control patients (Arm 3). PFS is defined as the time between first vaccination and first documentation of either disease progression/recurrence, or death without prior progression/recurrence.
Time Frame: From date of first vaccine until time disease progression or death without prior progression/recurrence, up to 48 months
Population: Progression free survival in patients receiving vaccine vs placebo.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Plus pp65-flLAMP DC With GM-CSF and Td (Arm 2): Given under the skin at day 22-24 after the first temozolomide cycle then at 2 week intervals. Doses 4-10 will be given on day 22-24 of each temozolomide cycle. Doses will continue until a total of 10 or until progression or unacceptable toxicity.
  pp65-shLAMP DC with GM-CSF (Arm 1) pp65-flLAMP DC with GM-CSF (Arm 2)
  Td: All subjects will receive a Td booster before study drug dose #1. Subjects in the experimental arms will receive Td skin prep before study drug doses #3, #6, and #9.
Arm/Group | pp65-shLAMP DC With GM-CSF and Td (Arm 1) | Plus pp65-flLAMP DC With GM-CSF and Td (Arm 2) | Unpulsed PBMC and Saline (Arm 3)
Number analyzed (Participants) | 36 | 34 | 41
months | 6.1 [3.9 to 11.0] | 6.4 [4.2 to 10.8] | 7.1 [3.9 to 14.8]
Statistical Analysis 1: Comparison: pp65-shLAMP DC With GM-CSF and Td (Arm 1) vs Unpulsed PBMC and Saline (Arm 3); Test type: Superiority; p = 0.354, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.60 to 1.61]
Statistical Analysis 2: Comparison: Plus pp65-flLAMP DC With GM-CSF and Td (Arm 2) vs Unpulsed PBMC and Saline (Arm 3); Test type: Superiority; p = 0.354, Log Rank; Hazard Ratio (HR) = 1.42, 95% CI 2-sided [0.87 to 2.33]

3. Secondary Outcome: ELISPOT Assay (pp65)
Description: Within patient changes from baseline to vaccine 3.
Time Frame: baseline, post-vaccine #3
Population: Participants in each arm who received at least 3 DC vaccines.
Measure: Mean (Standard Deviation); unit: spot forming units (SFU)
Groups:
- Arm 1: pp65-shLAMP DC With GM-CSF and Td: Given under the skin at day 22-24 after the first temozolomide cycle then at 2 week intervals. Doses 4-10 will be given on day 22-24 of each temozolomide cycle. Doses will continue until a total of 10 or until progression or unacceptable toxicity.
  pp65-shLAMP DC with GM-CSF
  Td: All subjects will receive a Td booster before study drug dose #1. Subjects in the experimental arms will receive Td skin prep before study drug doses #3, #6, and #9.
- Arm 2: pp65-flLAMP DC With GM-CSF and Td: Given under the skin at day 22-24 after the first temozolomide cycle then at 2 week intervals. Doses 4-10 will be given on day 22-24 of each temozolomide cycle. Doses will continue until a total of 10 or until progression or unacceptable toxicity.
  Td: All subjects will receive a Td booster before study drug dose #1. Subjects in the experimental arms will receive Td skin prep before study drug doses #3, #6, and #9.
  pp65-flLAMP DC with GM-CSF
- Arm 3: Unpulsed PBMC and Saline: Given under the skin at day 22-24 after the first temozolomide cycle then at 2 week intervals. Doses 4-10 will be given on day 22-24 of each temozolomide cycle. Doses will continue until a total of 10 or until progression or unacceptable toxicity.
  unpulsed PBMC and saline
  Saline
Arm/Group | Arm 1: pp65-shLAMP DC With GM-CSF and Td | Arm 2: pp65-flLAMP DC With GM-CSF and Td | Arm 3: Unpulsed PBMC and Saline
Number analyzed (Participants) | 20 | 26 | 29
spot forming units (SFU) | 126.3 (759.9) | 48.4 (377.5) | -162.7 (1075.4)
Statistical Analysis 1: Comparison: Arm 1: pp65-shLAMP DC With GM-CSF and Td; Test type: Superiority; p = 0.038, Kruskal-Wallis
Statistical Analysis 2: Comparison: Arm 2: pp65-flLAMP DC With GM-CSF and Td; Test type: Superiority; p = 0.038, Kruskal-Wallis
Statistical Analysis 3: Comparison: Arm 3: Unpulsed PBMC and Saline; Test type: Superiority; p = 0.038, Kruskal-Wallis

4. Secondary Outcome: Flow Cytometric Analysis (T Cell)
Description: Percentage of circulating cellular subsets of T cells within PBMCs.
Time Frame: baseline, post-vaccine #3
Population: Only participants who received at least 3 DC vaccines are included.
Measure: Mean (Standard Deviation); unit: percentage of PBMC
Groups:
- pp65-shLAMP DC With GM-CSF and Td (Arm 1); pp65-flLAMP DC With GM-CSF and Td (Arm 2): Prior to leukapheresis, patients will be randomized to receive one of three treatment regimens with dose-intensified TMZ treatment at 100 mg/m2/day for 21 days with an allocation ratio of 1:1:1 into one of three arms.
  DC vaccines are given under the skin at day 22-24 after the first temozolomide cycle then at 2-week intervals. Doses 4-10 will be given on day 22-24 of each temozolomide cycle. Doses will continue until a total of 10 or until progression or unacceptable toxicity.
  Td: All subjects will receive a Td booster before study drug dose #1. Subjects in the experimental arms will receive Td skin prep before study drug doses #3, #6, and #9.
Arm/Group | pp65-shLAMP DC With GM-CSF and Td (Arm 1) | pp65-flLAMP DC With GM-CSF and Td (Arm 2) | Unpulsed PBMC and Saline (Arm 3)
Number analyzed (Participants) | 15 | 19 | 17
percentage of PBMC | -0.1 (11.1) | 5.9 (16.6) | 1.7 (7.0)

5. Secondary Outcome: Cytokine Array Analysis (IFN-g)
Description: Change in concentration (pg/mL) of IFN-g as measured by multiplex array from Baseline (V1) to post-Vaccine #3.
Time Frame: baseline, post-vaccine #3
Population: Only participants who received at least 3 DC vaccines are included in the analysis
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | pp65-shLAMP DC With GM-CSF and Td (Arm 1) | pp65-flLAMP DC With GM-CSF and Td (Arm 2) | Unpulsed PBMC and Saline (Arm 3)
Number analyzed (Participants) | 25 | 30 | 33
pg/mL | -3.5 (5.0) | 3.3 (17.7) | -1.7 (10.0)
Statistical Analysis 1: Comparison: pp65-shLAMP DC With GM-CSF and Td (Arm 1); Test type: Superiority; p = 0.2, Kruskal-Wallis
Statistical Analysis 2: Comparison: pp65-flLAMP DC With GM-CSF and Td (Arm 2); Test type: Superiority; p = 0.2, Kruskal-Wallis
Statistical Analysis 3: Comparison: Unpulsed PBMC and Saline (Arm 3); Test type: Superiority; p = 0.2, Kruskal-Wallis

6. Secondary Outcome: ELISPOT Assay (Actin)
Description: Within patient changes from baseline to vaccine 3.
Time Frame: baseline, post-vaccine #3
Population: Participants in each arm who received at least 3 DC vaccines.
Measure: Mean (Standard Deviation); unit: spot forming units (SFU)
Arm/Group | Arm 1: pp65-shLAMP DC With GM-CSF and Td | Arm 2: pp65-flLAMP DC With GM-CSF and Td | Arm 3: Unpulsed PBMC and Saline
Number analyzed (Participants) | 20 | 26 | 29
spot forming units (SFU) | 0.4 (6.0) | -0.2 (26.1) | -0.4 (9.4)
Statistical Analysis 1: Comparison: Arm 1: pp65-shLAMP DC With GM-CSF and Td; Test type: Superiority; p = 0.6, Kruskal-Wallis
Statistical Analysis 2: Comparison: Arm 2: pp65-flLAMP DC With GM-CSF and Td; Test type: Superiority; p = 0.6, Kruskal-Wallis
Statistical Analysis 3: Comparison: Arm 3: Unpulsed PBMC and Saline; Test type: Other; p = 0.6, Kruskal-Wallis

7. Secondary Outcome: Flow Cytometric Analysis (NK Cell)
Description: Percentage of circulating cellular subsets of NK cells within PBMCs.
Time Frame: baseline, post-vaccine #3
Population: Only participants who received at least 3 DC vaccines are included.
Measure: Mean (Standard Deviation); unit: percentage of PBMC
Arm/Group | pp65-shLAMP DC With GM-CSF and Td (Arm 1) | pp65-flLAMP DC With GM-CSF and Td (Arm 2) | Unpulsed PBMC and Saline (Arm 3)
Number analyzed (Participants) | 15 | 19 | 17
percentage of PBMC | -1.3 (11.1) | 5.9 (16.6) | 1.7 (7.0)

8. Secondary Outcome: Flow Cytometric Analysis (CD4.CD25 T Reg)
Description: Percentage of circulating cellular subsets of CD4.CD25 T Reg within PBMCs.
Time Frame: baseline, post-vaccine #3
Population: Only participants who received at least 3 DC vaccines are included.
Measure: Mean (Standard Deviation); unit: percentage of PBMC
Arm/Group | pp65-shLAMP DC With GM-CSF and Td (Arm 1) | pp65-flLAMP DC With GM-CSF and Td (Arm 2) | Unpulsed PBMC and Saline (Arm 3)
Number analyzed (Participants) | 15 | 19 | 17
percentage of PBMC | -0.1 (4.3) | 1.4 (2.2) | -0.1 (2.0)
Statistical Analysis 1: Comparison: pp65-shLAMP DC With GM-CSF and Td (Arm 1); Test type: Superiority; p = 0.13, Kruskal-Wallis
Statistical Analysis 2: Comparison: pp65-flLAMP DC With GM-CSF and Td (Arm 2); Test type: Superiority; p = 0.13, Kruskal-Wallis
Statistical Analysis 3: Comparison: Unpulsed PBMC and Saline (Arm 3); Test type: Superiority; p = 0.13, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: AE collection began at the time of administration of vaccine #1 and continued until 30 days after the last dose of study drug, up to 13 months for each participant. All-cause mortality was assessed up to 48 months.
Description: The reporting of Adverse Events is based on the efficacy analysis set (mITT), which includes all subjects who receive at least one DC vaccine. 111 participants were included in modified intent to treat; for purposes of AE reporting, the N was 110 after we excluded 1 participant who did not meet AE reporting criteria.
Groups:
- pp65-shLAMP DC With GM-CSF and Td (Arm 1); pp65-flLAMP DC With GM-CSF and Td (Arm 2): The active treatment group was arms 1 and 2 combined.
  Arm 1: pp65-shLAMP mRNA DCs with GM-CSF 150 µg (Td skin prep) Arm 2: pp65-flLAMP mRNA DCs with GM-CSF 150 µg (Td skin prep)
Arm/Group | pp65-shLAMP DC With GM-CSF and Td (Arm 1) | pp65-flLAMP DC With GM-CSF and Td (Arm 2) | Unpulsed PBMC and Saline (Arm 3)
All-Cause Mortality (participants affected / at risk) | 28/36 | 31/34 | 31/41
Serious Adverse Events (participants affected / at risk) | 8/36 | 6/34 | 5/41
Other Adverse Events (participants affected / at risk) | 16/36 | 11/34 | 13/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | pp65-shLAMP DC With GM-CSF and Td (Arm 1) (N=36) | pp65-flLAMP DC With GM-CSF and Td (Arm 2) (N=34) | Unpulsed PBMC and Saline (Arm 3) (N=41)
Bruising (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Gastrointestinal - Other (Specify, appendicitis) (Gastrointestinal disorders) | 0 | 1 | 0
Hematoma (Blood and lymphatic system disorders) | 0 | 1 | 0
Infection (Infections and infestations) | 2 | 1 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 | 0 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Neurology - Other (Specify, cerebral edema) (Nervous system disorders) | 3 | 2 | 1
Seizure (Nervous system disorders) | 4 | 1 | 0
Syncope (fainting) (Nervous system disorders) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | pp65-shLAMP DC With GM-CSF and Td (Arm 1) (N=36) | pp65-flLAMP DC With GM-CSF and Td (Arm 2) (N=34) | Unpulsed PBMC and Saline (Arm 3) (N=41)
CD4 Count (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 4 | 6 | 5
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 1 | 0 | 0
Platelets (Blood and lymphatic system disorders) | 1 | 2 | 2
Hypertension (Cardiac disorders) | 2 | 0 | 4
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 | 1 | 0
Bruising (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0
Gastrointestinal - Other (Gastrointestinal disorders) | 0 | 1 | 0
Hematoma (Blood and lymphatic system disorders) | 0 | 1 | 0
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 | 0 | 0
Infection - Other (Infections and infestations) | 1 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Kidney (Infections and infestations) | 0 | 0 | 1
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 1 | 1 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 | 1 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 | 0 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Mood alteration - Depression (Nervous system disorders) | 1 | 0 | 0
Neurology - Other (Nervous system disorders) | 4 | 2 | 3
Pyramidal tract dysfunction (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 5 | 3 | 1
Syncope (fainting) (Nervous system disorders) | 0 | 1 | 0
Pain - Head/headache (General disorders) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT02465268/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT02465268/ICF_000.pdf